CLINICAL TRIAL: NCT00337077
Title: A Phase II Trial of E7389 (Halichondrin B Analog), in Patients With Metastatic Hormone Refractory Prostate Cancer
Brief Title: Eribulin Mesylate in Treating Patients With Metastatic Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00566; NCI-2009-00566 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E5805 (Other: Eastern Cooperative Oncology Group (ECOG)); U10CA021115 (NIH)
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Results first posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-04

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-refractory Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
Keywords: Eribulin Mesylate; metastatic hormone refractory prostate cancer; Halichondrin B Analog
MeSH Terms: conditions — Prostatic Neoplasms | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eribulin mesylate (Experimental): Patients receive eribulin mesylate IV over 5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: eribulin mesylate

INTERVENTIONS:
Drug: eribulin mesylate — Given IV
  Other Names: B1939; E7389; ER-086526; halichrondrin B analog

SUMMARY:
This phase II trial is studying how well eribulin mesylate (E7389; Halichondrin B Analog) works in treating patients with metastatic prostate cancer that did not respond to hormone therapy. Drugs used in chemotherapy, such as eribulin mesylate, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the number of patients with a > 50% decrease in prostate-specific antigen (PSA) of at least 4 weeks duration in patients with hormone-refractory metastatic prostate cancer treated with E7389 (eribulin mesylate).

SECONDARY OBJECTIVES:

I. Estimate the measurable disease response in patients with measurable disease.

II. Determine the duration of PSA and measurable disease response.

III. Characterize the safety and tolerability of E7389 in these patients.

OUTLINE:

This study enrolled 3 cohorts of patients based on the number of prior chemotherapy regimens received. The 3 cohorts are chemonaive stratum, prior-taxane stratum, and two-prior-chemotherapy stratum. Patients receive eribulin mesylate intravenously (IV) over 5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate
* Progressive metastatic disease or stable metastatic disease with rising PSA
* Previously treated with bilateral orchiectomy or other primary hormonal therapy with evidence of treatment failure
* Patients who have not undergone bilateral orchiectomy must continue luteinizing hormone-releasing hormone (LHRH)-agonist therapy (e.g., leuprolide or goserelin) or LHRH antagonist therapy (e.g. abarelix) while receiving study treatment
* Patients who did not have an orchiectomy must have a testosterone level < 50 ng/dL to confirm androgen suppression within the past 4 weeks
* ECOG performance status 0-2
* Adequate bone marrow function
* Bilirubin =< 1.5 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 times upper limit of normal
* Creatinine =< 2.0 mg/dL OR creatinine clearance >= 40 mL/min
* Fertile patients must use effective contraception
* A taxane-based regimen, mitoxantrone, or other cytotoxic chemotherapy regimen allowed provided there is evidence of disease progression
* At least 4 weeks since prior chemotherapy or radiotherapy
* At least 4 weeks since prior flutamide (6 weeks for bicalutamide or nilutamide) and there is continued evidence of disease progression
* Disease progression after antiandrogen withdrawal must be confirmed by rising PSA after the required 4-6 week washout period (e.g., PSA level higher than the last PSA obtained while on antiandrogen therapy)
* More than 4 weeks since prior estrogen, estrogen-like agents (e.g., PC-SPES, saw palmetto, or other herbal products that may contain phytoestrogens), or any other hormonal therapy (including megestrol, finasteride, ketoconazole, or systemic corticosteroids)
* Concurrent bisphosphonates (e.g., pamidronate sodium or zoledronate) allowed provided the patient has been receiving the bisphosphonate for >= 4 weeks and there is evidence of disease progression

Exclusion Criteria:

* Active angina pectoris
* Known New York Heart Association class III-IV heart disease
* Myocardial infarction within the past 6 months
* Evidence of ventricular dysrhythmias or other unstable arrhythmia (rate-controlled atrial fibrillation is allowed if the patient is asymptomatic from a cardiac standpoint)
* Peripheral neuropathy > grade 2
* Other prior malignancy (excluding nonmelanomatous skin cancer treated with curative intent) unless the malignancy was treated with curative intent and the patient has been disease free for >= 5 years
* Serious concurrent medical illness or active infection that would preclude study treatment - No concurrent strong inhibitors or inducers of CYP3A4
* More than 2 prior chemotherapy regimens for hormone-refractory disease - Other concurrent investigational agents
* Other concurrent anticancer therapy, including chemotherapy, gene therapy, biologic therapy, or immunotherapy
* Concurrent palliative radiotherapy
* Concurrent estrogen, estrogen-like agents, or any other hormonal therapy
* Carcinomatous meningitis or brain metastases
* Prior strontium chloride Sr 89, samarium 153 lexidronam pentasodium, or other radioisotopes
* Concurrent therapeutic anticoagulation with warfarin (Unfractionated heparin [standard, low-dose, or adjusted dose] or low molecular weight heparin allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-11; Primary Completion 2009-06 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stein, M.D., Study Chair — Rutgers Cancer Institute of New Jersey
Locations (147):
- United States (147):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Community Hospital of Monterey Peninsula, Monterey, California
  - Manchester Memorial Hospital, Manchester, Connecticut
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Evanston CCOP-NorthShore University HealthSystem, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Carle Foundation - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - Indiana University Health La Porte Hospital, La Porte, Indiana
  - Saint Anthony Memorial Health Center, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Eastern Cooperative Oncology Group, Boston, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hackensack University Medical CCOP, Hackensack, New Jersey
  - Cancer Institute of New Jersey At Hamilton, Hamilton, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - New York University Langone Medical Center, New York, New York
  - The North Division of Montefiore Medical Center, The Bronx, New York
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Cancer Center at Saint Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Saint Luke's Hospital, Bethlehem, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - UW Health Oncology - 1 South Park, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Riverview Hospital, Wisconsin Rapids, Wisconsin

REFERENCES:
- [Result] Stein MN, Chen Y, Hudes GR, Carducci MA, Tan W, DiPaola RS. ECOG 5805: A phase II study of eribulin mesylate (E7389) in patients (pts) with metastatic castration-resistant prostate cancer (CRPC). J Clin Oncol 28:15s, 2010 (suppl; abstr 4556)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from ECOG member institutions between November 29, 2006 and August 5, 2009.
Groups:
- Chemonaive: Patients who did not receive any prior chemotherapy. Patients receive eribulin mesylate intravenously (IV) over 5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Prior Taxane: Patients who received one prior taxane regimen. Patients receive eribulin mesylate intravenously (IV) over 5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Two Prior Chemotherapy Regimens: Patients who received two prior chemotherapy regimens. Patients receive eribulin mesylate intravenously (IV) over 5 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Chemonaive | Prior Taxane | Two Prior Chemotherapy Regimens
Started | 43 | 53 | 25
Treated | 42 | 52 | 25
Toxicity Assessed | 42 | 51 | 25
Eligible and Treated | 41 | 51 | 24
Patients With Measurable Disease | 26 | 38 | 13
Completed | 0 (No completion of treatment because treatment was given until PD or unacceptable toxicity.) | 0 (No completion of treatment because treatment was given until PD or unacceptable toxicity.) | 0 (No completion of treatment because treatment was given until PD or unacceptable toxicity.)
Not Completed | 43 | 53 | 25
Not completed — Progressive disease | 25 | 37 | 19
Not completed — Adverse Event | 7 | 7 | 1
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 7 | 2 | 2
Not completed — Alternative therapy | 1 | 0 | 0
Not completed — Physician Decision | 1 | 4 | 2
Not completed — Never started treatment | 1 | 1 | 0
Not completed — Ineligible | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients are included in this analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemonaive | Prior Taxane | Two Prior Chemotherapy Regimens | Total
Number analyzed (Participants) | 41 | 51 | 24 | 116
Age, Continuous [Median (Full Range); unit: years] | 70 [45 to 86] | 67 [45 to 88] | 73 [57 to 85] | 70 [45 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 41 | 51 | 24 | 116
Region of Enrollment [Number; unit: participants]
  United States | 41 | 51 | 24 | 116

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With PSA Response
Description: PSA response is defined as a PSA decline from baseline value by >=50%, or normalization of PSA (<0.2 ng/ml) confirmed by a second measurement greater than or equal to 4 weeks later.
Time Frame: Assessed every 3 weeks during treatment; after off-treatment, every 3 months if patient is <2 years from study entry and every 6 months if patient is 2-5 years
Population: Eligible and treated patients are included in this analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Chemonaive | Prior Taxane | Two Prior Chemotherapy Regimens
Number analyzed (Participants) | 41 | 51 | 24
Proportion of participants | 0.293 [0.182 to 0.442] | 0.098 [0.052 to 0.271] | 0.042 [0.004 to 0.152]

2. Secondary Outcome: Proportion of Patients With Measurable Disease Response
Description: Measurable disease response was evaluated using RECIST (Response Evaluation Criteria in Solid Tumors) 1.0 criteria. Per RECIST criteria, complete response (CR) = disappearance of all target and non-target lesions. Partial response (PR)= >=30% decrease in the sum of the longest diameters of target lesions from baseline, and persistence of one or more non-target lesion(s) and/or the maintenance of tumor marker level above the normal limits. Measurable disease response = CR + PR. Only patients with measurable disease at baseline are included in this analysis.
Time Frame: Assessed every 9 weeks during treatment; after off-treatment, every 3 months if patient is <2 years from study entry and every 6 months if patient is 2-5 years from study entry
Population: Eligible and treated patients with measurable disease at baseline are included in this analysis.
Measure: Number (90% Confidence Interval); unit: Proportion of participants
Arm/Group | Chemonaive | Prior Taxane | Two Prior Chemotherapy Regimens
Number analyzed (Participants) | 26 | 38 | 13
Proportion of participants | 0.154 [0.054 to 0.318] | 0.026 [0.001 to 0.119] | 0.077 [0.004 to 0.316]

ADVERSE EVENTS:
Time Frame: Assessed every 3 weeks while on treatment and for 30 days after the end of treatment
Groups:
- Eribulin Mesylate: All treated patients are evaluated for toxicities except for one patient who died soon after starting treatment and was not assessed for toxicity.
Arm/Group | Eribulin Mesylate
Serious Adverse Events (participants affected / at risk) | 81/118
Other Adverse Events (participants affected / at risk) | 111/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=118)
Anemia (Blood and lymphatic system disorders) | 9
Leukocytes decreased (Investigations) | 49
Lymphopenia (Investigations) | 3
Neutrophils decreased (Investigations) | 65
Hypotension (Vascular disorders) | 2
Fatigue (General disorders) | 13
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 3
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Bladder, hemorrhage (Renal and urinary disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 5
Infection w/ gr3-4 neut, sinus (Infections and infestations) | 1
Infection Gr0-2 neut, blood (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Extremity-lower (gait/walking) (General disorders) | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 2
Confusion (Psychiatric disorders) | 1
Neuropathy-motor (Nervous system disorders) | 3
Neuropathy-sensory (Nervous system disorders) | 15
Syncope (Nervous system disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 1
Pain-other (General disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=118)
Anemia (Blood and lymphatic system disorders) | 74
Leukocytes decreased (Investigations) | 74
Lymphopenia (Investigations) | 8
Neutrophils decreased (Investigations) | 56
Platelets decreased (Investigations) | 11
Hypotension (Vascular disorders) | 6
Fatigue (General disorders) | 82
Insomnia (Psychiatric disorders) | 6
Weight loss (Investigations) | 17
Alopecia (Skin and subcutaneous tissue disorders) | 46
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 38
Constipation (Gastrointestinal disorders) | 33
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 19
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 40
Taste disturbance (Nervous system disorders) | 11
Vomiting (Gastrointestinal disorders) | 9
Edema limb (General disorders) | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 22
Alkaline phosphatase increased (Investigations) | 14
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 11
Hypocalcemia (Metabolism and nutrition disorders) | 7
Creatinine increased (Investigations) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 15
Neuropathy-sensory (Nervous system disorders) | 45
Tearing (Eye disorders) | 6
Joint, pain (Musculoskeletal and connective tissue disorders) | 6
Muscle, pain (Musculoskeletal and connective tissue disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less